CLINICAL TRIAL: NCT00636727
Title: A Comparison of Arthrocentesis, Arthroscopy and Arthroplasty in the Treatment of Temporomandibular Joint Dysfunction
Acronym: TMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Gary F Bouloux MD, DDS, MDSc, FRACDS, FRACDS, Doctor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000450
Record Dates: First submitted 2008-02-15; First posted 2008-03-14 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: arthrocentesis; arthroscopy; arthroplasty
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthrocentesis; Arthroscopy; Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): arthrocentesis
  Interventions: Procedure: arthrocentesis
- 2 (Active Comparator): arthroscopy
  Interventions: Procedure: arthroscopy
- 3 (Active Comparator): arthroplasty
  Interventions: Procedure: arthroplasty

INTERVENTIONS:
Procedure: arthrocentesis — Irrigate the TMJ with lactated ringers
  Arms: 1
Procedure: arthroscopy — The TMJ will be inspected with an arthroscope and the joint irrigated with lactated ringers
  Arms: 2
Procedure: arthroplasty — The disc will be surgically repositioned with open surgery
  Arms: 3

SUMMARY:
Many patients suffer from a disorder known as temporomandibular joint dysfunction. This disorder has jaw joint pain and limited function as key elements. Many treatments have been advocated over the last 40 years, many of them deleterious. Currently treatment can be divided into four categories. The first is non-surgical and involves vocal rest, soft diet, heat, anti-inflammatory medications, muscle relaxants, splint therapy and physical therapy. All patients benefit to some degree utilizing one or more non-surgical approaches. Controversy exists with respect to which of the next three categories of treatment is ideal. Some advocate arthrocentesis which involves placing two small needles into the joint to allow irrigation and instillation of anti-inflammatory medication. This is a minimally invasive procedure performed under local anesthetic alone or with intravenous sedation. Others advocate arthroscopy which involves placing an arthroscope (a thin tube about 2mm in diameter with optical elements allowing one to see inside a joint) to visualize the inside of a joint. Furthermore the joint can be irrigated, scar bands removed, ligaments stretched and medication instilled. This is performed under a general anesthesia. Depending on the study, success for both arthrocentesis and arthroscopy has been reported to be about 80-90%. Still there are others who recommend arthroplasty which is an open joint surgical procedure that allows the surgeon to enter the joint and directly repair or remove the damaged cartilage disc within the joint. This is performed under a general anesthesia. Similar success rates of 80-94% have been reported. It is clear that some patients only require arthrocentesis, others arthroscopy and others arthroplasty. We currently do not have any real mechanism of predicting which patients will benefit the most from which procedure.

This study will enable patients undergoing each procedure to be followed closely with the hope that we can determine objective factors that will allow us to stratify patients into one of the three surgical options: arthrocentesis, arthroscopy or arthroplasty. Our current approach is empiric and typically proceeds from arthrocentesis to arthroscopy to arthroplasty. All patients in this study will be offered the opportunity to have arthrocentesis performed. It is anticipated that a minority will achieve long-term benefit in terms of pain and function. We hope to be able to identify those factors which will predict which patients will benefit so that future patients selected to have arthrocentesis will have much higher success rates. Patients who fail to improve with arthrocentesis or who initially decline that procedure will be offered the opportunity to undergo arthroscopy. It is anticipated that a majority of patients will achieve long-term benefit in terms of pain and function. Again it is hoped that we can identify those factors which will predict which patients will benefit so that future patients selected to have arthroscopy will have even higher success rates. Patients who fail to improve with arthroscopy or who initially decline both arthrocentesis and arthroscopy will be offered the opportunity to undergo arthroplasty provided that clinical and radiographic evidence exists to support the presence of either a diseased or displaced cartilage disc.

Our ability to adequately treat patients with temporomandibular joint dysfunction will be significantly improved if we can better stratify patients and follow an evidence based surgical algorithm that provides the greatest opportunity for success while reducing potential complications. Each of these surgical procedures is the standard of care throughout the USA but unfortunately the choice of which procedure to perform is often empiric and guided more by training and surgical experience.

ELIGIBILITY:
Inclusion Criteria:

* All patients who require a surgical intervention

Exclusion Criteria:

* None

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Reduction in pain | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary f Bouloux, MD, DDS, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States